CLINICAL TRIAL: NCT05268952
Title: A Prospective, Multicentric, Proof-of-concept Study to Evaluate the Value of Circulating Tumour DNA in Follow-up of Patients With an Advanced Gastroenteropancreatic or Lung Neuroendocrine Tumour Under Everolimus +- SSA Treatment
Brief Title: A Study to Evaluate the Value of Circulating Tumour DNA in Follow-up of Patients With an Advanced Gastroenteropancreatic or Lung Neuroendocrine Tumour Under Everolimus +- SSA Treatment (Liquid-NET 2.0)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Universiteit Antwerpen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Liquid-NET 2.0
Record Dates: First submitted 2022-01-21; First posted 2022-03-07 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-01

CONDITIONS: Neuroendocrine Tumors
Keywords: Liquid biopsies
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Liquid Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GEP-NET and lung-NET patients (Experimental): Liquid biopsies and scans
  Interventions: Other: Liquid biopsies; Other: Scans (CT, gallium-68 DOTATE/TOC/NOC PET-CT)

INTERVENTIONS:
Other: Liquid biopsies — Blood/urine sampling and scans are done at regular intervals
Other: Scans (CT, gallium-68 DOTATE/TOC/NOC PET-CT) — Scans will be done at regular intervals

SUMMARY:
Prospective, multicentric, single arm, POC study to evaluate the value of CtDNA in follow-up of patients treated with everolimus, with or without somatostatin analogues for advanced gastroenteropancreatic or lung neuroendocrine tumours.

DETAILED DESCRIPTION:
Prospective, multicentric, single arm, POC study to evaluate the value of CtDNA in follow-up of patients treated with everolimus, with or without somatostatin analogues for advanced gastroenteropancreatic or lung neuroendocrine tumours. Inclusion is possible after proven progressive disease on CT and/or DOTANOC scan (at physician's discretion) and decision of physician to start everolimus ± SSA treatment. During the study, CT and/or DOTANOC scans (thorax/abdomen/pelvis) (at physician's discretion) will be performed to detect progressive disease and CtDNA levels will be measured from the start of the treatment. The changes in CtDNA levels will be correlated to the tumour disease progression based on imaging (RECIST 1.1 and or PERCIST 1.0 (if available)) and laboratory and clinical markers. Characterization of CtDNA will be based on detection of tumour-specific alterations (i.e. mutations, copy number alterations and DNA methylation) using next-generation sequencing, digital droplet PCR and a photoelectrochemical biosensor. The identification of tumour-specific mutations will be done using next-generation sequencing of tumour tissue.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Written informed consent prior to any study-related procedure
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Histological proven diagnosis of a well or moderately differentiated GEP-NET (WHO2017 grade 1,2,3 neuroendocrine tumour)
* Documented progressive gastroenteropancreatic or lung neuroendocrine tumour by means of imaging and based upon the RECIST 1.1 criteria and/or PERCIST 1.0 criteria (if available) for which the treating physician has decided to treat with everolimus ± SSA treatment
* Presenting a positive CT and/or DOTANOC scan (at physician's discretion) at study entry with a measurable tumour lesion > 1 cm (CT scan with a maximum slice thickness of 5 mm); baseline CT and/or DOTANOC scan performed up to 28 days prior start of treatment NO previous treatment with everolimus
* Adequate bone marrow and coagulation function as shown by:

  1. Haemoglobin ≥ 9.0 g/dL
  2. ANC ≥ 1,500/mm3 (≥1.5 x 109/L)
  3. Platelets ≥ 100,000/mm3 (≥ 100x 109/L)
  4. INR ≤ 2.0
* Adequate liver function as shown by:

  1. Alanine aminotransferase and aspartate aminotransferase ≤2.5xULN (Upper limit of normal) (or ≤ 5 if hepatic metastases are present)
  2. Total serum bilirubin ≤ 1.5 x ULN (≤ 3 ULN for patients known to have Gilbert Syndrome)
* Adequate renal function as shown by Serum creatinine≤ 1.5 x ULN
* Fasting serum cholesterol, triglycerides and glucose

  1. Fasting serum cholesterol ≤ 300 mg/dL or 7.75 mmol/L
  2. Fasting triglycerides ≤ 2.5 x ULN
  3. Fasting glucose < 1.5 x ULN
* Availability of FFPE tissue of GEP-NET or lung NET tumour tissue or patient willing to have a new biopsy in case of non-availability of tissue

Exclusion Criteria:

* Patients with only non-measurable lesions by CT
* Known hypersensitivity to mTOR inhibitors, e.g. sirolimus (rapamycin) or other contra-indications for everolimus ± SSA treatment
* Unavailable archival tissue and patient unwilling to have a new biopsy
* Prior treatment with everolimus
* History of drug hypersensitivity with a similar chemical structure to lanreotide Autogel 120mg, sandostatin LAR or everolimus
* Unresolved Grade 3 or 4 toxicity from prior therapy, including experimental therapy
* History or clinical evidence of other malignancy within 3 years prior to enrolment, with the exception of adequately treated in-situ carcinoma of the cervix, uteri, basal or squamous cell carcinoma or non-melanomatous skin cancer
* Major surgery within 4 weeks of first dose administration
* History of symptomatic brain metastases or other central nervous system metastases.
* Patients receiving concomitant immunosuppressive agents or chronic corticosteroid use at the time of study entry except in cases outlined below:
* Topical applications (e.g. rash) Inhaled sprays (e.g. obstructive airways disease)
* Eye drops
* Local injections (e.g. intra-articular)
* Stable low dose of corticosteroids for at least two weeks before enrolment
* Patients with known HIV seropositivity. Screening for HIV infection at baseline is not required
* Acute and chronic, active infectious disorders (including hepatitis patients)
* Chronic pulmonary medical conditions or acute respiratory problems
* Active bleeding diathesis
* On oral anti-vitamin K medication with an INR ≥3
* Any severe uncontrolled medical condition such as:

  1. Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction ≤ 6 months prior to enrolment, uncontrolled cardiac arrhythmia
  2. Uncontrolled diabetes defined as fasting glycemia > 150 mg/dl.
  3. Acute and chronic, active infectious disorders and non-malignant medical illnesses that are uncontrolled or whose control may be jeopardized by the complications of this study therapy.
  4. Symptomatic deterioration of lung function
* Patients being treated with drugs recognized as being strong inhibitors or inducers of the isoenzyme CYP3A (Rifabutin, Rifampicin, Clarithromycin, Ketoconazole, Itraconazoleonazole, Voriconazole, Ritonavir, Telithromycin) within the last 5 days prior to enrolment
* Patients that will likely require treatment during the study with drugs that are not permitted by the study protocol.
* History of non-compliance to medical regimens
* Concurrent anti-cancer treatment in another investigational trial, other than the everolimus ± SSA treatment
* Patients that are likely to require any additional concomitant treatment with anti-proliferative effect for the pancreatic neuroendocrine tumour
* Patients unwilling or unable to comply with the protocol or patients with mental condition rendering the patient unable to understand the nature, scope and possible consequences of the study, and/or evidence of an uncooperative attitude
* Any abnormal findings at baseline, clinical finding, including psychiatric and behavioural problems, or any other medical condition(s) or laboratory findings that, in the opinion of the investigator, might jeopardize the patient's safety or decrease the chance of obtaining satisfactory data needed to achieve the objective(s) of the study
* Childbearing potential (unless using an adequate measure of contraception)
* Pregnancy or lactation. Females of childbearing potential must provide a negative pregnancy test at the start of study and must be using oral, double barrier or injectable contraception. Non-childbearing potential is defined as post-menopausal for at least 1 year, surgical sterilization or hysterectomy at least three months before the start of the study.
* Has previously been enrolled in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-05-27 (Actual); Primary Completion 2025-05-27 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of treatment follow-up through CtDNA level measurement | 48 months
  Feasibility of treatment follow-up through detection of a change in CtDNA levels before progression is apparent on imaging according to RECIST 1.1 and/or PERCIST 1.0 (if available) (Progression-free survival (PFS)).

SECONDARY OUTCOMES:
PFS under everolimus ± SSA treatment | 48 months
  PFS under everolimus ± SSA treatment
Overall response rates under everolimus ± SSA treatment | 48 months
  Overall response rates under everolimus ± SSA treatment
Safety of everolimus ± SSA treatment according to the Common Terminology Criteria for Adverse Events 4 (CTCAE4) and in Belgium according to the Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) | 48 months
  Number of patients with (serious) adverse events throughout the study
Comparison of PFS based on RECIST 1.1 and PERCIST 1.0 | 48 months
  Comparison of PFS based on RECIST 1.1 and PERCIST 1.0

CONTACTS AND LOCATIONS:
Locations (3):
- Belgium (2):
  - Antwerp University Hospital, Edegem, Antwerp
  - VITAZ, Sint-Niklaas, East-Flanders
- Bank of Cyprus Oncology Center, Nicosia, Cyprus

IPD SHARING:
Plan to Share IPD: No